CLINICAL TRIAL: NCT06890325
Title: A Service-Learning Program for Comprehensive Geriatric Assessment and Health Promotion in Older Adults
Acronym: GEROS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Javier Jerez Roig, Associate Professor, Head of the Research Group M3O, Care Area Coordinator of the IRIS-CC, University of Vic - Central University of Catalonia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24/082; 2023 IMPAC 00014 (Other Grant/Funding Number: AGAUR)
Record Dates: First submitted 2025-03-05; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Frailty; Older People; Comprehensive Geriatric Assessment; Health Promotion; SERVICE LEARNING; Students; Student Education
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Comprehensive geriatric assessment. (Experimental): Comprehensive geriatric assessment.
  Interventions: Diagnostic Test: Comprehensive Geriatric Assessment (CGA); Behavioral: Health education

INTERVENTIONS:
Diagnostic Test: Comprehensive Geriatric Assessment (CGA) — The intervention will consist of a total of 3 sessions which will take place in different areas of the Faculty of Health and Welfare Sciences (FCSB) at the University of Vic - Central University of Catalonia. In Session 1, a comprehensive geriatric assessment (CGA) will be conducted to the users (by students supervised by health professionals).
Behavioral: Health education — A report with the results of the CGA and health recommendations will be delivered to the users. They will receive health education including specific recommendations and community health resources based on their health status and CGGA.

SUMMARY:
The GEROS Project aims to develop and implement a Service-Learning (S-L) program that integrates Comprehensive Geriatric Assessment (CGA) and health promotion, for students at the Faculty of Health Sciences and Welfare at the University of Vic - Central University of Catalonia (UVic-UCC). This initiative engages university students, healthcare professionals, and older adults (60+) in a participatory, intergenerational approach that fosters mutual learning and community engagement.

The study follows a non-experimental mixed-method design, involving students from Nursing, Physiotherapy, Human Nutrition and Dietetics, Occupational Therapy, and Psychology. Participants include older adults (60+) who can independently travel to the university.

The project is integrated into different subjects, in groups of 4-5 students, participants conduct a Comprehensive Geriatric Assessment (CGA), evaluating frailty using VIG-Frail, intrinsic capacity with ICOPE, quality of life with EUROQOL 5D-5L, and specific health indicators with Nursing Outcomes Classification (NOC).

To assess the program's effectiveness, several outcome measures will be analyzed including students' perceived knowledge, competencies, and skills, as well as older adults' awareness of their health status, lifestyle, and risk factors. Additionally, the satisfaction levels of both will be evaluated. The items will be evaluated using a 1-5 Likert Scale, and the analysis will be conducted with SPSS. Data recording will be carried out through REDCap.

The GEROS Project aligns with the United Nations' Sustainable Development Goals (SDGs), specifically SDG 3 (Good Health and Well-being) and SDG 10 (Reduced Inequalities). By offering care to the aging population and providing them with personalized health recommendations, the project promotes preventive strategies, active aging, and intergenerational learning.

Furthermore, GEROS integrates innovative educational methodologies, encouraging experiential learning, collaboration with healthcare professionals, and the development of practical skills in real-world contexts. The program's scalability and adaptability could serve as a model for other universities and healthcare institutions aiming to enhance geriatric care through service-learning initiatives.

ELIGIBILITY:
Inclusion Criteria:

A) For users:

* Any person aged 60 or older who can move to the facility (Faculty of Health Sciences and Welfare) independently or accompanied by a caregiver.

B) For students:

* Students from Nursing, Physiotherapy, Nutrition and Dietetics, Occupational Therapy and Psychology degrees of UVic-UCC.

Exclusion Criteria:

* For users: Individuals institutionalized in a long-term care institution.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Frailty | Baseline assessment
  VIG-Frail is a screening tool used to assess frailty in older adults. It's a short, easy-to-administer test that helps healthcare providers identify individuals who may be at risk of adverse health outcomes due to frailty.
Users Satisfaction with treatment | Up to 2-4 weeks (Post-intervention - 2nd session)
  Evaluation of the user's general satisfaction with participating in the project (5-point Likert scale from 1-not at all to 5-very satisfied)
Students Satisfaction with intervention | At the end of Session 1 (CGA of users)
  Evaluation of the students' general satisfaction with the participation in the study (5-point Likert scale from 1-not at all to 5-very satisfied)

SECONDARY OUTCOMES:
Self-reported Quality of Life | Baseline assessment
  Quality of Life measured with EuroQol 5D-5L, a standardised tool used to measure and assess health-related quality of life. The "5D" refers to five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels, ranging from "no problems" to "extreme problems," allowing for a detailed assessment of a person's health status.Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as.
Intrinsic capacity | Baseline assessment
  Integrated care for older people approach (ICOPE) is a framework developed by the World Health Organization to support the health and well-being of older adults through comprehensive, integrated care.
  It focuses on 7 key dimensions: cognitive decline, limited mobility, undernutrition, vision impairment, hearing loss, depressive symptoms, and social care and supports, as well as carer support and urinary incontinence. These areas are assessed to create a holistic care plan tailored to the individual's needs. This outcome will be categorized according to the number or preserved dimensions: from 7 (all 7 dimesions preserved) to 0 (all 7 dimensions affected).
Nursing Outcomes Classification | Baseline assessment
  The NOC (Nursing Outcomes Classification) is a system used to assess the results of nursing care, helping to measure a person's level of functioning and well-being in different areas of health.
  The NOC outcomes evaluated in this context are: Cognition, Mobility, Nutritional Status, Sensory Function: Vision, Desire to Live, Caregiver Well-being Urinary Continence, Psychosocial Adjustment: Life Change These outcomes are assessed using a 5-point Likert scale, ranging from 1 (Not demonstrated) to 5 (Always demonstrated).
Students Self-perception of increased knowledge, skills and competencies | At the end of Session 1 (CGA of users)
  Knowledge about Health Promotion and Disease Prevention, Improvement in Skills and Technical Competencies in Comprehensive Geriatric Assessment (CGA), Skills and Technical Competencies in Intrinsic Capacity (ICOPE), Transversal Skill "Communication", Critical Thinking, Integration of Knowledge, Skills, and Competencies in the subject in Which the project Was Held, Problem-Solving Ability, Interdisciplinary. These outcomes are assessed using a 5-point Likert scale, ranging from 1 (Not demonstrated) to 5 (Always demonstrated).
Users Self-perception of increased knowledge, skills and competencies | Up to 2-4 weeks (Post-intervention - 2nd session)
  Knowledge about Their Own Health, Lifestyle and Risk Factors to Modify for increasing Health and Disease Prevention and Community Health Resources, evaluated with a Likert scale from 1 to 5 (1 = not much, 5 = very much)

CONTACTS AND LOCATIONS:
Overall Officials: Júlia Casacuberta-Roca, Nursing, Study Director — University of Vic - Central University of Catalonia
Locations (1):
- Faculty of Health Sciences and Welfare, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No